CLINICAL TRIAL: NCT02506257
Title: Randomized, Double-Masked, Placebo-Controlled Multiple-Dose Phase 1 Study to Evaluate the Safety and Tolerability of Different Doses of Preservative-free Polyhexamethylene Biguanide (PHMB) Ophthalmic Solution in Healthy Subjects
Brief Title: Safety and Tolerability of Preservative-free Polyhexamethylene Biguanide (PHMB) Ophthalmic Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 042SI
Record Dates: First submitted 2015-07-20; First posted 2015-07-23 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Acanthamoeba Keratitis
MeSH Terms: conditions — Acanthamoeba Keratitis | interventions — polihexanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.04% PHMB (Experimental): 0.04% PHMB eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Interventions: Drug: 0.04% PHMB
- 0.06% PHMB (Experimental): 0.06% PHMB eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Interventions: Drug: 0.06% PHMB
- 0.08% PHMB (Experimental): 0.08% PHMB eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Interventions: Drug: 0.08% PHMB
- PHMB Vehicle (Placebo Comparator): PHMB vehicle eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Interventions: Drug: PHMB Vehicle

INTERVENTIONS:
Drug: 0.04% PHMB — 0.04% PHMB eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Other Names: Polyhexamethylene Biguanide
  Arms: 0.04% PHMB
Drug: 0.06% PHMB — 0.06% PHMB eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Other Names: Polyhexamethylene Biguanide
  Arms: 0.06% PHMB
Drug: 0.08% PHMB — 0.08% PHMB eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Other Names: Polyhexamethylene Biguanide
  Arms: 0.08% PHMB
Drug: PHMB Vehicle — PHMB vehicle eye drops, 1 drop 12 times daily for 7 days, followed by 1 drop 6 times daily for additional 7 days
  Arms: PHMB Vehicle

SUMMARY:
Randomized, double-masked, placebo-controlled, multiple center, parallel-group Phase 1 study to evaluate the safety and tolerability of 3 doses of preservative-free PHMB ophthalmic solution compared to placebo in healthy subjects

DETAILED DESCRIPTION:
The primary objective of the study is to establish the ocular safety and tolerability, and systemic safety of 3 different concentrations of preservative-free PHMB in healthy subjects. Safety and tolerability will be compared to those of a placebo.The PHMB bioavailability in plasma will also be assessed

ELIGIBILITY:
Inclusion Criteria:

* able and willing to give informed consent.
* man or woman of any race and 18 to 55 years of age, inclusive.
* Body Mass Index of 20-30 kg/m2
* willing and able to attend required study visits.
* bilateral visual acuity >6/10.
* intraocular pressure (IOP) of 14-21 mmHg.
* ophthalmologic examination without abnormalities.
* medical history without major pathology.
* laboratory test results without deviations from the normal range.
* female subjects of childbearing potential with negative urine pregnancy test and using effective contraception during the study.

Exclusion Criteria:

* presence of bacterial ocular infections.
* presence of any concomitant ocular pathology.
* performing activities likely to result in an irritated conjunctiva during the study (including heavy alcohol intake, swimming in chlorinated water and heavy smoking).
* contact lenses wearing .
* ocular surface fluorescein staining score >3.
* use of topical or systemic antibiotics, antihistamines, decongestants and non-steroidal anti-inflammatory agents as well as steroids within 7 days before screening.
* known or suspected allergy to biguanides or intolerance to any other ingredient of the test treatments.
* ocular surgery performed within 12 months before screening.
* participation in another clinical study in the preceding 30 days.
* one functional eye.
* pregnancy or breastfeeding.
* use of recreational drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I JE van der meulen, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papa V, van der Meulen I, Rottey S, Sallet G, Overweel J, Asero N, Minassian DC, Dart JKG. Safety and tolerability of topical polyhexamethylene biguanide: a randomised clinical trial in healthy adult volunteers. Br J Ophthalmol. 2022 Feb;106(2):190-196. doi: 10.1136/bjophthalmol-2020-317848. Epub 2020 Nov 25. PMID 33239413

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Started | 26 | 28 | 27 | 9
Completed | 26 | 26 | 23 | 9
Not Completed | 0 | 2 | 4 | 0
Not completed — Adverse Event | 0 | 2 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Adult healthy volunteers
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle | Total
Number analyzed (Participants) | 26 | 28 | 27 | 9 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (12.5) | 29.4 (8.7) | 30.4 (10.3) | 25.7 (4.6) | 29.6 (10.1)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 15 | 17 | 2 | 48
  Male | 12 | 13 | 10 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose-limiting Adverse Events
Time Frame: up to 21 days from date of randomization
Measure: Number; unit: participants
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Number analyzed (Participants) | 26 | 28 | 27 | 9
participants | 0 | 2 | 3 | 0

2. Secondary Outcome: Plasma Concentration of PHMB
Time Frame: Day14
Measure: Mean (Standard Deviation); unit: micrograms/ml
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Number analyzed (Participants) | 26 | 28 | 27 | 9
micrograms/ml | 0 (0) | 0 (0) | 0 (0) | 0 (0)

3. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Change from baseline systolic blood pressure
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Number analyzed (Participants) | 26 | 28 | 27 | 9
mmHg | -0.7 (9.6) | 0.6 (8.3) | -0.9 (8.6) | 1.0 (8.6)

4. Other Pre Specified Outcome: Visual Acuity
Description: Change from baseline Visual acuity. Best corrected visual acuity was reported in decimal fraction. A decrease of visual acuity during treatment was considered a negative safety outcome.
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: decimals
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Number analyzed (Participants) | 26 | 28 | 27 | 9
decimals | 0.3 (1.4) | 0.3 (1.3) | 0.3 (0.1) | 0.3 (0.1)

5. Other Pre Specified Outcome: Ocular Surface Disease Index-OSDI
Description: Change from baseline OSDI at D 14. Score range was betwwen 0-100. An increase of OSDI values with treatment represent a negative outcome.
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Number analyzed (Participants) | 26 | 28 | 27 | 9
scores on a scale | 1.5 (3.6) | 1.3 (4.1) | 4.2 (5.8) | -2.2 (4.9)

6. Other Pre Specified Outcome: Conjunctival Examination
Description: Change from baseline conjunctival staining at Day 14. Staining with lissamine green was used. The density of staining was graded with the Oxford Score. Score range was between 0-15. An increase in the score after treatment represent a negative outcome
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Number analyzed (Participants) | 26 | 28 | 27 | 9
scores on a scale | 0.7 (1.3) | 1.2 (1.9) | 1.7 (1.8) | 1.0 (1.7)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | 0.04% PHMB | 0.06% PHMB | 0.08% PHMB | PHMB Vehicle
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28 | 0/27 | 0/9
Other Adverse Events (participants affected / at risk) | 11/26 | 23/28 | 16/27 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.04% PHMB (N=26) | 0.06% PHMB (N=28) | 0.08% PHMB (N=27) | PHMB Vehicle (N=9)
conjunctival hypermia (Eye disorders) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Instillation site pain (General disorders) | 2 (2) | 4 (4) | 5 (5) | 1 (1)
conjunctival staining (Investigations) | 2 (3) | 5 (5) | 9 (11) | 0 (0)
corneal staining (Investigations) | 1 (1) | 5 (5) | 8 (8) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 4 (5) | 1 (1) | 1 (9)
eyelid edema (Eye disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Instillation site pain erythema (General disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Instillation site pruritus (General disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Instillation site foreign body sensation (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No